CLINICAL TRIAL: NCT01184950
Title: Prospective Randomized Trial of Virtual Reality Simulator Training in an Obstetrics and Gynecology Residency
Brief Title: Virtual Reality Laparoscopy Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Devin Namaky, MD, TriHealth Department of Obstetrics and Gynecology
Purpose: Other
Other Study IDs: 10019
Record Dates: First submitted 2010-08-11; First posted 2010-08-19 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2010-08

CONDITIONS: Differences in OSATS Scores

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trainer Curriculum (Experimental)
  Interventions: Other: Trainer Curriculum
- No Curriculum (No Intervention)

INTERVENTIONS:
Other: Trainer Curriculum
  Arms: Trainer Curriculum

SUMMARY:
The use of virtual reality simulation training in obstetrics and gynecology has not been widely studied. The investigators hypothesized that residents randomized to the trainer would not perform differently when compared with those who are not randomized. Residents in Obstetrics and gynecology are randomized to a 4 month training course on our simulator. They are objectively evaluated performing various laparoscopy tasks prior to and after the course.

ELIGIBILITY:
Inclusion Criteria:

* Resident in OB/Gyn at TriHealth

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
observed structured assessment of technical skills (OSATS) Score | 0 Months
  The residents are timed in seconds on various laparoscopy tasks. They are also rated by an objective blinded observer in several performance categories and given a score by the observer. These times and scores are recorded upon entry into the study, after randomization to intervention or no intervention.

SECONDARY OUTCOMES:
observed structured assessment of technical skills (OSATS) score | 4 Months
  The residents are timed in seconds on various laparoscopy tasks. They are also rated by an objective blinded observer in several performance categories and given a score by the observer. These times and scores are recorded 4 months after entry into the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States